CLINICAL TRIAL: NCT04900519
Title: A Phase 1, Open-Label, Dose-Escalation Study of the Safety and Efficacy of STI-6643, an Anti-CD47 Human Monoclonal Antibody, in Subjects With Advanced Solid Tumors
Brief Title: Study of the Safety and Efficacy of STI-6643 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47MAB-ADVCA-101
Record Dates: First submitted 2021-05-17; First posted 2021-05-25 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor; Relapsed Solid Neoplasm; Refractory Tumor
Keywords: solid tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- STI-6643 (Experimental): STI-6643 will be provided in a single use 10-mL high borosilicate type 1 glass vial at a concentration of 500mg/10 mL (50 mg/mL) administered intravenously weekly for 4 weeks, then biweekly for Cycles 2 and up.
  Interventions: Biological: STI-6643

INTERVENTIONS:
Biological: STI-6643 — Anti-CD47 human monoclonal antibody

SUMMARY:
This is a first-in-human, phase 1, open-label, dose-escalation study of STI-6643 administered by intravenous infusion in subjects with a relapsed/refractory advanced solid tumor.

DETAILED DESCRIPTION:
This is a first-in-human, phase 1, open-label, dose-escalation study of STI-6643 administered by intravenous infusion in subjects with a relapsed/refractory advanced solid tumor.

The study will determine an MTD and RP2D using a conventional 3+3 study design with priming dose identification (PDI) stage and therapeutic dose (TD) escalation (TDE) stage. Dose limiting toxicity evaluated over the initial 28 days of STI-6643 administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age ≥ 18 years
* ECOG Performance Status ≤ 2
* Histologically- or cytologically-confirmed solid tumor
* Patient has relapsed, is refractory to, or intolerant of standard of care therapy
* No available approved therapy that may provide clinical benefit (per Investigator)
* Measurable or evaluable disease by RECISTv1.14
* Life expectancy of > 12 weeks (per Investigator)
* Adequate laboratory parameters including:

  1. Absolute neutrophil count (ANC) ≥ 1500/mm3
  2. Platelets ≥ 100,000/mm3
  3. Hemoglobin ≥ 12 g/dL (in the absence of transfusion over the prior 2 weeks)
  4. AST/SGOT ≤ 2.5 x ULN (≤ 5 x ULN if known liver involvement)
  5. ALT/SGPT ≤ 2.5 x ULN (≤ 5 x ULN if known liver involvement)
  6. Total bilirubin ≤ 2.0 x ULN (unless diagnosis of Gilbert's syndrome in which case < 3.0 times ULN)
  7. Serum creatinine ≤ 2.0 x ULN or estimated GFR ≥ 45 mL/min (per Cockcroft- Gault equation)
* If residual treatment related toxicity from prior therapy:

  1. Treatment related toxicity resolved to ≤ Grade 1 (alopecia excepted), or
  2. Treatment related toxicity resolved to ≤ Grade 2 with prior approval of the Medical Monitor
* Willingness to comply with the study schedule and all study requirements
* [Females] Must be postmenopausal, surgically sterile, or agree to use adequate contraception (per Investigator) throughout the study and for a least 30 days following the last dose
* [Males] Must be surgically sterile or must agree to use adequate contraception (per Investigator) throughout the study and for at least 30 days following the last dose
* [Males] Willingness to refrain from donating sperm throughout the study and for at least 30 days following the last dose
* [Females] If of child-bearing potential, must have a negative serum pregnancy test

Exclusion Criteria:

* Participating in any other interventional clinical study
* Previous exposure to an anti-CD47 or SIRPα antibody
* ≤ 28 days (or 5 half-lives if shorter) between of systemic anti-tumor treatment (e.g., chemotherapy, endocrine therapy, immunotherapy, cellular therapy) and the 1st dose of STI-6643
* ≤ 28 days from prior irradiation (≤ 7 days from limited field irradiation for control of symptoms) and the 1st dose of STI-6643
* ≤ 28 days between major surgery (≤ 7 days from minor surgical procedures, no waiting period following central catheter placement)
* ≤ 7 days between administration of G-CSF, GM-CSF, erythropoietin, thrombopoietin or IL11 and the 1st dose of STI-6643
* ≤ 7 days between systemic immunosuppressive therapy in excess of 10 mg/day prednisone equivalent and the 1st dose of STI-6643 (topical or inhaled corticosteroids not restricted)
* ≤ 28 days between a live attenuated vaccine and the 1st dose of STI-6643
* Known central nervous system (CNS) involvement with tumor (e.g., metastases, meningeal carcinomatosis)
* Active second malignancy requiring ongoing systemic treatment
* History of primary immunodeficiency disorders
* History of active pulmonary tuberculosis
* History of COVID-19 symptoms unless COVID-19 test negative ≤ 72 hours of the 1st dose of STI-6643
* ≤ 12 weeks from an allogeneic hematopoietic stem cell transplant and C1D1 or active graft-versus-host disease (GvHD)
* Active infection (e.g., bacterial, viral, fungal) requiring systemic treatment ≤ 72 hours of the 1st dose of STI-6643
* Known HIV-positive with CD4+ cell counts < 350 cells/uL or a history of an AIDS defining opportunistic infection
* Known T-cell leukemia virus type 1 (HTLV1) infection, hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia
* Significant risk for HBV reactivation (defined as HbsAg positive, HbcAb positive or HBV DNA positive)
* Detectable HCV RNA
* Pregnant or breast feeding
* History of clinically significant cardiovascular abnormalities including:

  1. Congestive heart failure (NYHA classification ≥ 3) within 6 months of the 1st dose of STI-6643
  2. Unstable angina pectoris
  3. ≤ 6 months from myocardial infarction and the 1st dose of STI-6643
  4. Arrhythmias (other than atrial fibrillation) requiring ongoing treatment
  5. QTcF interval > 480 msec (using Fridericia's formula)
  6. Uncontrolled hypertension (i.e., systolic BP > 180 mmHg or diastolic BP > 100
* Any condition, including the presence of laboratory abnormalities, that places the subject at an unacceptable risk if the subject was to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-24 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Safety of STI-6643 | Baseline through study completion at up to approximately 31 months
  Safety as assessed by incidence of adverse events, SAEs, DLTs, and clinically significant changes in safety lab results

SECONDARY OUTCOMES:
Overall response rate | Day 1 through study completion at up to approximately 31 months
  Overall response rate
Duration of response | Day 1 through study completion at up to approximately 31 months
  Duration of response
STI-6643 receptor occupancy | Day 1 through Day 22
  STI-6643 receptor occupancy
Anti-drug antibodies directed to STI-6643 | Day 1 through Day 15
  Anti-drug antibodies directed to STI-6643
PK parameters | Day 1 through Day 22
  Evaluate the pharmacokinetics of STI-6643

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (5):
- United States (5):
  - University of California, San Diego, San Diego, California
  - Sanford Health, Sioux Falls, South Dakota
  - NEXT Oncology - Austin, Austin, Texas
  - Mary Crowley Cancer Research, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia